CLINICAL TRIAL: NCT02132780
Title: The Impact of Autonomic Dysfunction on Liver-Related Symptoms in Non-Alcoholic Fatty Liver Disease and Their Relationship to Systemic Inflammation and Insulin Resistance
Brief Title: Autonomic Dysfunction in Non-Alcoholic Fatty Liver Disease
Acronym: AD-NAFLD
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM20000329; UL1TR000058 (NIH)
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Non-alcoholic Fatty Liver Disease; NAFLD; Fatty Liver, Nonalcoholic; Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
There is a significant association between autonomic dysfunction and symptoms experienced by NAFLD patients mediated by increased systemic inflammation and insulin resistance, resulting in deteriorating quality of life of affected patients; fatigue and other symptoms drive worsening autonomic dysfunction in these patients. We aim to describe the severity of autonomic dysfunction (AD) in non-alcoholic fatty liver disease (NAFLD) and the relationship of AD to symptoms experienced by NAFLD patients (such as fatigue, chronic pain, depression, sleep disturbance, and cognitive dysfunction), and to the quality of life of NAFLD patients. We also hope to examine the impact of systemic inflammation and insulin resistance as mediators of manifestations of AD and symptoms experienced by NAFLD patients.

DETAILED DESCRIPTION:
Aim 1. Describe the severity of AD in NAFLD and the relationship of AD to symptoms experienced by NAFLD patients (fatigue, chronic pain, depression, sleep disturbance, and cognitive dysfunction) (Aim 1a) and to the quality of life of NAFLD patients (Aim 1b). Primary screening for inclusion/exclusion criteria will be done at the VCUHS clinic. Subjects meeting inclusion criteria will be approached about study participation during their routine NAFLD clinic visit. Those who agree to participate in the study will return for a study visit at the CCTR Clinical Research Services. All subjects will be asked to fast and avoid caffeine for 12 hours prior to study visit. Demographic and clinical data will be collected by study coordinators. After a focused exam, conducted by a hepatologist to determine health status of the participants, the PI and a research nurse will interview participants to assess their symptoms and AD (Aim 1). Blood (20 ml) samples will be collected via venipuncture for serum and plasma inflammatory markers and IR (Aim 2).

Aim 2. Examine the impact of systemic inflammation (SI) and insulin resistance (IR) as mediators of manifestations of AD and symptoms experienced by NAFLD patients. Increased presence of adipocytes may produce high, chronic levels of cytokines such as IL-6 and TNF-α resulting in higher levels of APRPs which contribute to overall inflammation as well as cognitive decline and fatigue. Secondly, elevated levels of IL-6 and TNF-α lower levels of CTRPs which exacerbate IR, AD, and muscle and cardiac problems reported in NAFLD. Through the use of plasma analysis, levels of cytokines such as IL-6, TNF-α, and APRPs can be performed in a high throughput BioPlex® assay (Bio-Rad Laboratories, Inc.: Hercules, CA). We have extensive experience with these types of assays and have generated data using human samples in numerous studies conducted through the Center of Excellence for Biobehavioral Approaches to Symptom Management (CEBASM) at the School of Nursing. CTRP family members are also expressed in the plasma and at detectible levels. We will perform ELISA analysis to compare circulating levels of the various CTRPs using commercially available CTRP ELISA kits/reagents. Insulin resistance (IR) will be assessed by HOMO-IR utilizing fasting glucose and insulin.

ELIGIBILITY:
Inclusion Criteria:

* Men and women within the age of 35-65
* understand and speak English
* NAFLD on liver histology by the biopsy within preceding 24 months

Exclusion Criteria:

* Patients with poorly controlled diabetes (HbA1c>8.5% or fasting blood glucose>150 mg/dl)
* renal dysfunction (Cr>1.5) last 3 months
* history of cardiac rhythm other than sinus rhythm
* on beta-blockers
* other liver diseases (HCV, HBV)
* decompensated cirrhosis (free of ascites hepatic encephalopathy, variceal bleeding)
* major depression
* cancer
* stroke
* any other major health conditions

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with NAFLD who are patients at the NAFLD Clinic at VCU Health Systems in Richmond, VA.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Autonomic Dysfunction | baseline
  Will record heart rate variability at the time of study visit and collect data from 24 hour automatic blood pressure readings. The Autonomic Symptoms Checklist will also be used.

SECONDARY OUTCOMES:
Relationship between AD and symptoms | baseline
  Data on symptoms will be collected using the Chronic Liver Disease Questionnaire and PROMIS symptom short forms for symptoms including fatigue, anxiety, sleep and depression. RBANS and Stroop will be used to assess cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Kyungeh An, PhD, Principal Investigator — VCU
Locations (1):
- Virginia Commonwealth University Health System, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
We completed this pilot with 23 participants. Sharing data is to be determined.